CLINICAL TRIAL: NCT02212912
Title: Cluster-randomized Trial of a Targeted Multifaceted Intervention to Bridge the Evidence-based Gap in the Management of Acute Ischemic Stroke
Brief Title: Intervention to Bridge the Evidence-based Gap in Stroke Care Quality
Acronym: GoldenBridge
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Yongjun Wang, Executive Vice-President, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: aic2014
Record Dates: First submitted 2014-08-02; First posted 2014-08-08 (Estimated); Last update posted 2020-07-13 (Actual); Status verified 2020-07

CONDITIONS: Ischemic Stroke
Keywords: acute ischemic stroke, performance measure, acute treatment
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Improvement intervention (Other): Improvement intervention is a multifaceted quality improvement method including evidence-based clinical pathway, standard operating procedures (SOP) of performance indicators, a quality coordinator, and monitoring and feedback system of performance measures.
  Interventions: Behavioral: improvement intervention
- no intervention (Other): The control group indicated that the physicians will not be provided with the information of multifacet improvement tools including evidence-based clinical pathway, standard operating procedures (SOP) of performance indicators a quality coordinator, and monitoring and feedback system of performance measures. They just provide patients with routine care
  Interventions: Behavioral: no intervention

INTERVENTIONS:
Behavioral: improvement intervention — Evidence-based clinical pathway: It contained general guideline-based recommendations about acute stroke management. Standard operating procedures (SOP) of performance indicators. A quality coordinator:The role of the quality coordinator includes interacting with physicians once gaps in the incorporation of evidence-based interventions are identified, ensuring that all components of the quality improvement intervention are being used for every acute ischemic stroke (AIS) patient.Monitoring and feedback system of performance measures.
  The system could view the level of implementation of prespecified performance measures at any time (per week recommended) , compare with the previous record of own study site and level of other clusters.
  Arms: Improvement intervention
Behavioral: no intervention — No intervention indicated that the physicians among control hospital provide routine
  Arms: no intervention

SUMMARY:
The purpose of this study is to evaluate whether a multifaceted quality improvement intervention can improve the adherent rate of individual and composite of evidence-based performance measures for patients with acute ischemic stroke within the first 7 days of symptom onset and reduce the incidence of a new clinical vascular event, disability, and all-cause mortality at discharge and long term clinical outcome.

DETAILED DESCRIPTION:
Study population:

patients with acute ischemic stroke who were admitted to the hospital within 7 days after the initial symptom onset.

Program:

There are multifaceted quality improvement interventions including:

1. Evidence-based clinical pathway
2. Standard operating procedures (SOP) of performance indicators
3. A quality coordinator
4. Monitoring and feedback system of performance measures

Endpoints:

Primary outcome:increase of adherence of evidence based treatment in clinical practice; Secondary outcome: total mortality, disability, and major cerebrovascular events

ELIGIBILITY:
Inclusion criteria:

* Older than 18
* Ischemic stroke within 7 days of the index event
* Direct admission based on physician evaluation or arrival through the emergency department
* Ability of patient or legally authorized representative to provide informed consent for 3, 6,and 12 months after initial symptom onset
* Eligible events were confirmed by brain ct or mri within7 days after the onset of symptoms

Exclusion criteria:

* Patients refuse to participate in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4800 (Actual)
Dates: Start 2014-08-10 (Actual); Primary Completion 2015-06-20 (Actual); Study Completion 2016-07-30 (Actual)

PRIMARY OUTCOMES:
percentage of all-or-none measure of evidence-based performance measures in acute ischemic stroke patients without contraindications | participants will be followed for the duration of hospital stay, an expected average of 2 weeks
  The primary end point was all-or-none measure of evidence-based performance measures in patients without contraindications, at the emergency department (Intravenous tissue-type plasminogen activator (tPA) in patients who arrive within 2 hours after initial symptom onset and treated within 3 hours), during 48 hours after admission (antithrombotic drugs; dysphagia screening; deep venous thrombosis prophylaxis including pneumatic compression devices, subcutaneous unfractionated heparin, low molecular weight heparin, or full-dose anticoagulation (e.g., with heparin or warfarin)) , and at discharge (antithrombotic therapy, discharge on anticoagulation for patients with atrial fibrillation, and discharged on statin, antihypertensive, and hypoglycemic medications). An all-or-none measure of care was used, which is defined as the proportion of patients who received all of the performance measure interventions for which they were eligible.
a composite measure score of performance measures | participants will be followed for the duration of hospital stay, an expected average of 2 weeks
  a composite measure score, defined as the total number of interventions performed among eligible patients divided by the total number of possible interventions among eligible patients, were also calculated.

SECONDARY OUTCOMES:
percentage of new clinical vascular event (ischemic stroke, hemorrhagic stroke, myocardial infarction, or vascular death) , disability (disability defined as Modified Rankin Score (mRS) ≥ 2) , and all-cause mortality | 3,6,12 months
  The secondary primary end point was a new clinical vascular event (ischemic stroke, hemorrhagic stroke, myocardial infarction, or vascular death) , disability (disability defined as Modified Rankin Score (mRS) ≥ 2) , and all-cause mortality at discharge,3, 6, 12-months after initial symptom onset.

OTHER OUTCOMES:
a composite measure score of performance measures | participants will be followed for the duration of hospital stay, an expected average of 2 weeks
  a composite measure score, defined as the total number of interventions performed among eligible patients divided by the total number of possible interventions among eligible patients, were also calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Yilong Wang, M.D, Principal Investigator — Beijing Tian Tan Hospital, Capital Medical University, Beijing, China; Yongjun Wang, M.D, Principal Investigator — Beijing Tian Tan Hospital, Capital Medical University, Beijing, China
Locations (1):
- Beijing Tian Tan Hospital, Capital Medical University, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Lynch EA, Bulto LN, Cheng H, Craig L, Luker JA, Bagot KL, Thayabaranathan T, Janssen H, McInnes E, Middleton S, Cadilhac DA. Interventions for the uptake of evidence-based recommendations in acute stroke settings. Cochrane Database Syst Rev. 2023 Aug 11;8(8):CD012520. doi: 10.1002/14651858.CD012520.pub2. PMID 37565934
- [Derived] Wang Y, Li Z, Zhao X, Wang C, Wang X, Wang D, Liang L, Liu L, Wang C, Li H, Shen H, Bettger J, Pan Y, Jiang Y, Yang X, Zhang C, Han X, Meng X, Yang X, Kang H, Yuan W, Fonarow GC, Peterson ED, Schwamm LH, Xian Y, Wang Y; GOLDEN BRIDGE-AIS Investigators. Effect of a Multifaceted Quality Improvement Intervention on Hospital Personnel Adherence to Performance Measures in Patients With Acute Ischemic Stroke in China: A Randomized Clinical Trial. JAMA. 2018 Jul 17;320(3):245-254. doi: 10.1001/jama.2018.8802. PMID 29959443
- [Derived] Wang Y, Li Z, Xian Y, Zhao X, Li H, Shen H, Wang C, Liu L, Wang C, Pan Y, Wang D, Prvu Bettger J, Fonarow GC, Schwamm LH, Smith SC Jr, Peterson ED, Wang Y; GOLDEN BRIDGE-AIS investigators. Rationale and design of a cluster-randomized multifaceted intervention trial to improve stroke care quality in China: The GOLDEN BRIDGE-Acute Ischemic Stroke. Am Heart J. 2015 Jun;169(6):767-774.e2. doi: 10.1016/j.ahj.2015.03.008. Epub 2015 Mar 26. PMID 26027613